CLINICAL TRIAL: NCT00814853
Title: Electrical Activity of the Diaphragm During Extubation Readiness Testing
Acronym: NAVA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Gerhard Wolf, MD - Instructor, Children's Hospital Boston, Harvard Medical School
Other Study IDs: 08-07-0338; ERT
Record Dates: First submitted 2008-12-24; First posted 2008-12-25 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Extubation
Keywords: Extubation; testing; ventilator weaning; Pediatric extubation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Extubation readiness testing: Patients who pass the ERT.
  Interventions: Device: NAVA (Extubation readiness testing failures)

INTERVENTIONS:
Device: NAVA (Extubation readiness testing failures) — Patients who fail the ERT will be place in the mode of ventilation NAVA.

SUMMARY:
Neurally adjusted ventilatory assist (NAVA) is a FDA approved mode of mechanical ventilation. This mode of ventilation is currently in routine use in adult, pediatric and neonatal intensive care units. The electrical activity of the diaphragm, the largest muscle used during respiration, is measured. The ventilator applies support in proportion to the measured electrical activity of the diaphragm (Edi). This electrical activity is measured through a feeding tube that also has a multiple-array esophageal electrode in it.

Whenever a patient gets extubated in our MSICU, we conduct a routine extubation readiness test. This is standard of care in our ICU. If the patient fails this test, the patient stays on the ventilator. If he passes, he gets extubated. We wish to conduct a study during which we will monitor the electrical activity of the diaphragm during this test. If the patient passes the extubation readiness test, the study is complete. If he fails, he resumes on the ventilator. In our study, we would then use the measured signal of the diaphragm to guide the ventilator. This mode of ventilation is called NAVA. We do not currently use this mode of ventilation in the ICU, but could do so since it is FDA approved. However, we wish to use this protocol to gain more expertise with this mode of ventilation in the ICU in a controlled fashion. We wish to enroll 20 pediatric patients. Patients in the ICU are routinely on a variety of different models of ventilators. Usually, the respiratory therapist determines which ventilator will be used. All patients in this study would be on the Servo-I ventilator, which is an FDA approved ventilator and capable of monitoring electrical activity of the diaphragm and currently used in our MSICU.

DETAILED DESCRIPTION:
1. Specific Aims /Objectives Specific Aim 1: To determine if Edi is a predictor of extubation readiness. (Hypothesis: an increase of 20-50% in Edi from baseline (prior to ERT) will predict successful extubation.) Specific Aim 2: If the patient fails the ERT - We hope to determine if NAVA will provide more information about why the patient failed the ERT. (Hypothesis: a decrease in peak inspiratory pressure from baseline (post ERT failure) is predictive of high frequency diaphragm fatigue and subsequent successful ERT.
2. Background and Significance The diaphragmatic function plays a pivotal role in the patient's ability to breathe on a ventilator, and on the successfulness of weaning from a ventilator and extubation. However, diaphragmatic function is not routinely measured in the ICU, which we would like to do in this trial.

   When the mechanical load of the respiratory system is too large or continues for a long period of time, the diaphragm can develop contractile fatigue[1]. This fatigue can be short or long term. Short term is also known as high-frequency fatigue that results from the accumulation of inorganic phosphate[2][3], and to a lesser extent intramuscular acidosis[4]. On the other hand long term fatigue, otherwise known as low-frequency fatigue is consistent with muscle injury[5, 6] and can persist for days. Being able to identify what type of diaphragm fatigue is present could help us understand the patient's readiness to be extubated.

   Despite the frequent use of mechanical ventilation, determining when to appropriately discontinue mechanical ventilation and extubate a patient remains a challenge. Many weaning protocols exist but are typically extrapolated from adult studies. These protocols can consist of but are not limited to use sprint weaning utilizing a T-piece (no support, just oxygen), continuous positive airway pressure (CPAP) or pressure support (PSV) trail. Usually, data is gathered through spirometry with a ventilator (shallow breathing index, tidal volumes, etc.) and vital signs are recorded [7, 8]. Despite the use of protocols extubation failure range from 15-24% (Randolph) in the pediatric population.

   Investigators have explored physiological evidence of improving lung function to help determine the appropriate time to discontinue mechanical ventilation. One notable effort by Hubble et al was to obtain dead space to tidal volume ratio (Vd/Vt) to determine extubation success after a 30 minute PSV trail prior to extubation[9]. They concluded that a Vd/Vt ratio of less than or equal to 0.5 reliably predicted successful extubation (96%). However, this only provides one part of the equation - lung function- but not necessarily the central nervous system interaction or the work of breathing associated.

   Currently, the MSICU uses an extubation readiness test (ERT). This test determines if patients are eligible for discontinuation of mechanical ventilation. This test consist of a daily screen of changing the FIO2 (fraction of inspired oxygen) to 50% (left at current setting if lower than 50%) and decrease the PEEP to 5 cmH2O. Patients unable to maintain saturation (SpO2) of 95%, or become tachypneic, or appear uncomfortable failed the test; those who maintained SpO2 of 95% or higher have their mode of ventilation changed to minimal pressure support (PSV). Minimal PSV was determined by the endotracheal tube (ETT) size. Patients were classified as failing the test if at any time in the two hour period their SpO2 was less than 95%, their exhaled tidal volume was less than 5 mL/kg ideal body weight, or their respiratory rate was outside of the acceptable range for age. If the patient fails an ERT they are returned to their previous ventilator setting and evaluated for extubation readiness in 24 hours. It is understood that sedation is one of the primary caused of extubation failure, however there is additional concern regarding the diaphragmatic function. When the mechanical load of the respiratory system is too large or continues for a long period of time, the diaphragm can develop contractile fatigue[4]. This fatigue can be short or long term. Short term is also known as high-frequency fatigue that results from the accumulation of inorganic phosphate[5], failure of the membrane electrical potential[6], and to a lesser extent intramuscular acidosis[7], but recover quickly. On the other hand long term fatigue, otherwise known as low-frequency fatigue is consistent with muscle injury [8, 9] and can persist for days. Being able to identify what type of diaphragm fatigue could lead us to hold on extubation readiness testing as to not re-injury.

   When patients are extubated too early, respiratory failure can occur [10, 11]. When extubation is delayed, lengths of time on mechanical ventilation and in the ICU stay both increases. This leads to additional respiratory complications such as ventilator associated pneumonia and overall lung damage[12]. Thus, the decision to extubate should be made on the basis of accurate, objective and reproducible criteria. The diaphragmatic activity is likely one of those criteria that are not yet measured. We aim to add some additional information to this body of knowledge that may link the respiratory pump (diaphragm) to lung function, muscle fatigue, and/or central nervous system depression.
3. Preliminary Studies/Progress Report To our knowledge there is not previous data determining if Edi can predict extubation success. However, there are a few limited studies on low and high-frequency diaphragm fatigue in adults and animals. Dr. Laghi and colleagues carefully examined 11 who failed extubation and eight adults whom successfully weaned from mechanical ventilation. They concluded that weaning itself did not cause low-frequency fatigue [13]. While Edi was examined in six health adults at high frequency fatigue levels. Edi was found to successfully assess neural drive and that diaphragm fatigue did not affect respiratory drive.

   Limits to the studies mentioned above that we plan to address are: none were done in children with highly resistive endotracheal tubes, length of mechanical ventilation was not examined (low vs. high frequency diaphragm fatigue risk), there was no formal ERT, and examination of low and high frequency diaphragm fatigue in the same patient population was not done.
4. Design and Methods a. Study Design In a prospective, blinded (Edi information blinded to the team) clinical trail we will study the diaphragmatic activity that occur prior and following our standard extubation readiness test (minimum pressure support trial). We will examine that diaphragmatic activity by examining the Edi prior to, during, and post the trial on every patient who qualifies. Furthermore, patients who fail ERT will be ventilated with the NAVA mode of ventilation. The entire protocol will be conducted on the Maquet Servo I ventilator

ELIGIBILITY:
Inclusion Criteria:

* All intubated and mechanically ventilated patients age 1 month to 18 years and meeting the extubation readiness criterion.

Exclusion Criteria:

* Patients in which a nasal gastric or oral gastric tube is contraindicated. Examples are but not limited to: s/p esophagus, tracheal surgery, bleeding disorders, facial trauma.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Anyone eligible for and extubation readiness test.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-12 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
EDI pre and post extubation readiness testing. | 2 hours

SECONDARY OUTCOMES:
Will the mode of ventilation NAVA wean the patient back to ERT settings. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Wolf, MD, Principal Investigator — Children's Hospital Boston, Harvard Medical School; Brian K Walsh, BS, RRT-NPS, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States